CLINICAL TRIAL: NCT06583122
Title: Ultrasound Guided Radiofrequency Ablation of the Occipital Nerve
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Timothy Sowder, MD, Principal Investigator, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00148697
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-12

CONDITIONS: Nerve Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ultrasound Guided Approach (Experimental): Ultrasound-guided approach to occipital nerve radiofrequency ablation
  Interventions: Procedure: Ultrasound Guided Approach

INTERVENTIONS:
Procedure: Ultrasound Guided Approach — All enrolled patients will receive the new ultrasound-guided approach to occipital nerve radiofrequency ablation

SUMMARY:
Study an ultrasound guided approach to radiofrequency ablation of the occipital nerve that makes it possible to see the needle during treatment procedure. It is hoped this will reduce the amount of pain after the standard of care procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-80 with a diagnosis of occipital neuralgia or migraine overlying the occipital region.
* A diagnosis of occipital neuralgia will be based on the International Classification of Headache Disorders (ICHD), whose criteria include: paroxysmal stabbing pain in the distribution of the GON, tenderness over the affected nerve, and relief of pain for at least 3 hours after bupivacaine local anesthetic block of the affected nerve.
* Patients may also be included if they have a diagnosis of migraine based on the ICHD criteria with predominance of pain over the occipital region that responded to occipital nerve block.
* Patients must have failed oral medications including NSAIDs, opioids, and anticonvulsants for the management of their pain.
* Failed treatment will be <50% pain reduction with oral medication.
* Patients must report headache frequency of at least 10 days per month.

Exclusion Criteria:

* Patients will be excluded from the trial if they have an unstable medical or psychological condition,
* are pregnant,
* have an implanted cardiac pacemaker or defibrillator that could not be disabled,
* have had a craniotomy or scar tissue overlying the site from a previous surgery,
* have a history of cervical spine fusion,
* have evidence of elevated ICP or intracranial tumor,
* or have previous RFA treatment of the greater or lesser occipital nerve.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction pain scores reported using an 11-point numeric rating scale (NRS) | 18 Months
  Pain scores will be assessed 0-10 at the beginning of the study and at the end. We will compare mean pain scores pre-intervention and post-intervention, and we expect mean pain scores will decrease by 4 points on the NRS

SECONDARY OUTCOMES:
Frequency of headache days | 18 months
  We will compare frequency of headache days pre-intervention and post-intervention
Frequency of moderate-severe headaches | 18 months
  We will compare frequency of moderate-severe headaches days pre-intervention and post-intervention
Use of acute pain medications | 18 Months
  We will compare frequency of Use of acute pain medications pre-intervention and post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No